CLINICAL TRIAL: NCT02693938
Title: Investigating Blood Glucose Variability and Insulin Action During Menstrual Cycle in Females With Type 1 Diabetes to Design Innovative Therapies
Brief Title: Blood Glucose Variability and Insulin Action During Menstrual Cycle in Females With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1509016531
Record Dates: First submitted 2016-01-15; First posted 2016-02-29 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; menstrual cycle; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- luteal phase clamp (Experimental): Luteal euglycemic clamp administered during luteal phase of menstrual cycle.
  Interventions: Device: Luteal Euglycemic clamp
- follicular phase clamp (Active Comparator): Follicular euglycemic clamp administered during follicular phase of menstrual cycle.
  Interventions: Device: Follicular Euglycemic clamp

INTERVENTIONS:
Device: Follicular Euglycemic clamp — Follicular Euglycemic clamp during follicular phase
  Arms: follicular phase clamp
Device: Luteal Euglycemic clamp — Luteal Euglycemic clamp during luteal phase
  Arms: luteal phase clamp

SUMMARY:
This research study is designed to look at differences in responsiveness to the subcutaneous injection of a standardized dose of rapid-acting insulin analog and blood glucose variability during different phases of the menstrual cycle in females with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
Type 1 Diabetes (T1D) is a chronic disease that leads to disability and premature death if not well treated. While females and males are equally affected by T1D, diabetes places additional burdens of care on females. Characteristically, females with T1D have worse glycemic control, a higher incidence of diabetic ketoacidosis, and a greater risk of cardiovascular complications as compared to their male peers. It has been hypothesized that variations in responsiveness to pre-meal bolus doses of insulin during menstrual cycling is an important underlying cause for increased management problems in females with T1D, but the hypothesis has not been adequately tested. Consequently, insulin treatment of females during the different cycles of menstruation remains a guessing game that often results in major swings in blood glucose from high to low levels. The unfavorable impact of this gap in knowledge extends to the efficiency and accuracy of artificial pancreas closed-loop (CL) system insulin delivery algorithms designed based on insulin action parameters. The proposed study addresses this unmet need in diabetes management for females both in open-loop (OL) and CL therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-35
2. diagnosis of T1D>1year;
3. BMI%<85th;
4. HbA1c <9%.
5. Subjects ages 21-35y on combination oral contraceptive pills (OCP) could be included.

Exclusion Criteria:

1. irregular periods,
2. pregnant, breastfeeding,
3. subjects>20y on progesterone only pills or injections,
4. Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol,
5. mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, including blood glucose monitoring requirements including the documentation of blood glucose data and insulin dosing,and/or inability to return for follow-up visits, and unlikely to complete the study.
6. Subjects on OCP will be excluded in the 12-20y group to capture the physiologic variability in insulin action during pubertal progress.

Ages: 12 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
The change in area under the glucose infusion rate (AUCGIR) during different phases of menstrual cycle | Up to 30 days
  The insulin glucodynamic action will be measured by the amount of dextrose infused during the study as previously described by DeFronzo. The primary outcome measure for the euglycemic clamp studies will be area under the glucose infusion rate (AUCGIR) that will be compared between luteal and follicular phases of menstrual cycle.
Glucose Infusion Rate | Up to 15 days
  During the luteal phase of the menstrual cycle, subjects will go through an insulin time action (clamp) study. Subjects are injected a bolus dose of insulin and blood sugar levels are kept within a 90-100mg/dL range by intravenous fluid infusion during fasting state. GIR stands for the glucose infusion rate that is measured in mg/kg/minute, indicating the amount of glucose delivered per minute per kilogram of body mass.
Glucose Infusion Rate | Up to 15 days
  During the follicular phase of the menstrual cycle, subjects will go through an insulin time action (clamp) study. Subjects are injected a bolus dose of insulin and blood sugar levels are kept within a 90-100mg/dL range by intravenous fluid infusion during fasting state. GIR stands for the glucose infusion rate that is measured in mg/kg/minute, indicating the amount of glucose delivered per minute per kilogram of body mass.

OTHER OUTCOMES:
Glycemic variability | Up to 30 days
  Glycemic variability measured by Continuous Glucose Monitor during two different phases of menstrual cycle will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Cengiz, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz C JL, Fabris C, Breton MD, Cengiz E. Insulin Replacement Across the Menstrual Cycle in Women with Type 1 Diabetes: An In Silico Assessment of the Need for Ad Hoc Technology. Diabetes Technol Ther. 2022 Nov;24(11):832-841. doi: 10.1089/dia.2022.0154. PMID 35714349